CLINICAL TRIAL: NCT03495869
Title: NIDA Phenotyping Assessments Battery (PhAB) Feasibility and Validation Study in Non-Intoxicated Drug Users
Brief Title: Feasibility and Validation of a Standard Phenotyping Assessment Battery
Acronym: PhAB
Status: Completed | Type: Observational
Sponsor: Virginia Commonwealth University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Other Study IDs: HM20012559; U54DA038999 (NIH)
Record Dates: First submitted 2018-03-29; First posted 2018-04-12 (Actual); Results first posted 2021-08-04 (Actual); Last update posted 2021-08-04 (Actual); Status verified 2021-07

CONDITIONS: Opioid-use Disorder; Cocaine Use Disorder; Marijuana Use Disorder; Healthy Controls
MeSH Terms: conditions — Opioid-Related Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- Individuals with Cocaine Use Disorder: This group will consist of individuals who are determined to have DSM5 diagnosis of Cocaine Use Disorder (n=50).
  Individuals will be recruited from an existing registry (VCU IRB HMHM20000294, Keyser-Marcus, PI)
- Individuals with Opioid Use Disorder: This group will consist of individuals who are determined to have DSM5 diagnosis of Opioid Use Disorder (n=200).
- Individuals with Marijuana Use Disorder: This group will consist of individuals who are determined to have DSM5 diagnosis of Marijuana Use Disorder (n=50).
- Healthy Controls: This group will consist of individuals who are determined to be non-drug using healthy controls (n=100).

SUMMARY:
The overall goal of this project is to collect preliminary data on psychosocial measures and behavioral performance comparing individuals with Opioid Use Disorder, Cocaine Use Disorder, dual diagnosis of Opioid and Cocaine Use Disorder, and Healthy Controls in an effort to determine overall feasibility of a phenotypic "fingerprint" for cohorts of individuals with addictions for use during clinical trials.

DETAILED DESCRIPTION:
There is profound heterogeneity of subjects in clinical studies of addictions, with patients being diagnosed by the primary substance of use. As a result, utilizing current DSM addictions classification leads to problems with signal detection and hamper the progress of the development of new drugs and treatments for substance use disorders (SUDs). Getting beyond the DSM-5 based definitions is necessary to "fingerprint" addiction phenotypes and endophenotypes, using machine-learning analyses of big data. A detailed in-depth assessment of addiction phenotypes (deep phenotyping) may also include neuroimaging.

In an effort to develop a "fingerprint" for addiction phenotypes, NIDA established a Workgroup to develop a phenotyping battery of tests and self-rated psychometric scales, supplemented by resting state fMRI to be administered to participants in any extramural clinical trial where addictions are assessed. The final phenotyping battery content was determined via consensus from both the selected experts- consultants group and the NIDA workgroup, and as such, the battery requires feasibility and validation study to finalize its content. The NIDA Phenotyping Assessment Battery (PhAB) covers six neurofunctional addiction domains: Metacognition, Interoception, Cognition/Executive Function, Reward/Incentive Salience, Emotion/Negative Emotionality, and Sleep/Circadian Rhythm. The PhAB is meant to be administered during a Phenotyping visit - an extension of a screening visit in any clinical trial addictions protocol. In addition to the PhAB, the group also developed an ancillary set of measures to be administered in conjunction with the PhAB in any addictions clinical trial during the Phenotyping visit. The Platform Instruments include structured interviews, diagnostic measures (e.g., MINI), self report scales of symptom severity (e.g., ASRS-ADHD, VAS-Pain), trauma history (CTQ), computer-administered measures of intelligence (e.g., Shipley), and substance use measures (FTND, Timeline Follow-back), etc. Clinical trial investigators would administer these scales and behavioral tasks in addition to protocol nonspecific assessments (e.g., demographics) and medical evaluations (e.g, medical history and physical exams, genotyping, and labs) which could be done at Screening.

This study is a feasibility, construct and face validity study. The primary outcome measure is time taken to complete the battery, and rates of successful study completion

ELIGIBILITY:
Inclusion Criteria (Individuals with SUDs)

* Males and females between 18 and 70 years-of-age.
* Current DSM-5 primary Substance Use Disorder: Opioid, marijuana, stimulants (individuals with multiple types of substance use (e.g., opioid/marijuana will be included)
* Have no contraindications for study participation as determined by medical history and concomitant medications.
* Be able to demonstrate an understanding of study procedures and follow instructions including behavioral laboratory testing.
* Be able and willing to comply with scheduled visits, and other study procedures.
* Be able to read and complete forms and interviews in English.

Inclusion Criteria (Non-drug Using Healthy Controls)

* Males and females between 18 and 70 years of age.
* Have no contraindications for study participation as determined by medical history and concomitant medications.
* Be able to demonstrate an understanding of study procedures and follow instructions including behavioral laboratory testing.
* Be able and willing to comply with scheduled visits, and other study
* Be able to read and complete forms and interviews in English.

General Exclusion Criteria

* Current psychosis, mania, or suicidal/homicidal ideation
* Meet current DSM-5 diagnosis of any psychoactive substance use disorder other than opioids,marijuana, stimulants, or nicotine. Diagnosis of mild to moderate use disorder for alcohol will not be considered exclusionary for any SUD group.
* Have a history of seizures (excluding childhood febrile seizures), or loss of consciousness from traumatic injury for more than 30 minutes.
* Have any other illness, or condition, which in the opinion of the PI or study physician would preclude safe and/or successful completion of the study.

MRI Exclusion Criteria

* Metal fragments or implants, and/or history of fear of being in closed spaces for MRI scans.
* Currently pregnant or nursing.

Ages: 18 Years to 70 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The study utilizes a four-group cross sectional cohort design. A total of 400 participants (across 4 cohorts) are targeted to complete the study) to include: Healthy Controls (n=100), individuals with CocUD (n=50), individuals with OUD (n=200), and individuals with MJUD (n=50).
Sampling Method: Non-Probability Sample
Enrollment: 368 (Actual)
Dates: Start 2018-06-21 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-03-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Keyser-Marcus, PhD, Principal Investigator — Virginia Commonwealth University
Locations (1):
- VCU Institute for Drug and Alcohol Studies, Richmond, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Individuals With Cocaine Use Disorder | Individuals With Opioid Use Disorder | Individuals With Marijuana Use Disorder | Healthy Controls
Started | 54 | 124 | 61 | 129
Completed | 50 | 97 | 51 | 108
Not Completed | 4 | 27 | 10 | 21
Not completed — Lost to Follow-up | 4 | 17 | 8 | 14
Not completed — Withdrawal by Subject | 0 | 3 | 0 | 3
Not completed — Dropped from study | 0 | 7 | 2 | 4

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Individuals With Cocaine Use Disorder | Individuals With Opioid Use Disorder | Individuals With Marijuana Use Disorder | Healthy Controls | Total
Number analyzed (Participants) | 50 | 97 | 51 | 108 | 306
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.78 (8.76) | 42.49 (11.57) | 35.24 (13.10) | 35.69 (14.51) | 40.77 (13.82)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 45 | 22 | 64 | 144
  Male | 37 | 52 | 29 | 44 | 162
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 2 | 1 | 3 | 7
  Not Hispanic or Latino | 44 | 91 | 46 | 99 | 280
  Unknown or Not Reported | 5 | 4 | 4 | 6 | 19
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: American Indian or Alaska Native | 0 | 0 | 1 | 4 | 5
  Race: Asian | 0 | 0 | 2 | 8 | 10
  Race: Native Hawaiian or Pacific Islander | 0 | 0 | 0 | 0 | 0
  Race: Black or African American | 48 | 72 | 31 | 42 | 193
  Race: White | 1 | 23 | 17 | 47 | 88
  Race: Other | 1 | 1 | 0 | 6 | 8
  Race: Unknown or not reported | 0 | 1 | 0 | 1 | 2
Region of Enrollment [Number; unit: participants]
  United States | 50 | 97 | 51 | 108 | 306

OUTCOME MEASURES:

1. Primary Outcome: Retention
Description: Number of dropouts
Time Frame: 1 month
Population: All participants who signed consent forms and screened eligible were included in the analysis for this outcome variable.
Measure: Count of Participants; unit: Participants
Arm/Group | Individuals With Cocaine Use Disorder | Individuals With Opioid Use Disorder | Individuals With Marijuana Use Disorder | Healthy Controls
Number analyzed (Participants) | 54 | 124 | 61 | 129
Participants | 4 | 27 | 10 | 21

2. Secondary Outcome: Time to Complete Battery
Description: Time to complete the assessment batteries will also be recorded for each task and each participant.
Time Frame: 5 hours
Measure: Mean (Standard Deviation); unit: Minutes
Arm/Group | Individuals With Cocaine Use Disorder | Individuals With Opioid Use Disorder | Individuals With Marijuana Use Disorder | Healthy Controls
Number analyzed (Participants) | 50 | 97 | 51 | 108
Minutes
  Time to complete Phenotyping assessment battery | 73.86 (15.77) | 68.53 (16.16) | 59.76 (10.19) | 61.04 (17.66)
  Time to complete battery of Platform Instruments | 96.97 (38.07) | 91.24 (32.83) | 75.08 (28.67) | 68.53 (24.52)

3. Secondary Outcome: Non-completers of the Battery and Platform Instruments
Description: Number of study completers who did not complete the full battery and platform instruments
Time Frame: 5 hours
Measure: Number; unit: participants
Arm/Group | Individuals With Cocaine Use Disorder | Individuals With Opioid Use Disorder | Individuals With Marijuana Use Disorder | Healthy Controls
Number analyzed (Participants) | 50 | 97 | 51 | 108
participants | 0 | 0 | 0 | 0

4. Other Pre Specified Outcome: Performance on Measures of Cognition Across Conditions
Description: Performance (time to complete)
  #correct) on behavioral tasks which examine cognitive functioning (e.g., Backwards digit span, and stop signal reaction task)
Time Frame: 5 hours
Reporting Status: Not Posted

5. Other Pre Specified Outcome: Performance on Measures of Reward Processing Across Conditions
Description: Performance (time to complete)
  #correct) on behavioral tasks which examine Reward processing (e.g., hypothetical purchase task) and subscale and total scale scores on self-report measures of reward processing (SUPP-S)
Time Frame: 5 hours
Reporting Status: Not Posted

6. Other Pre Specified Outcome: Performance on Measures of Negative Emotionality Across Conditions
Description: Performance (time to complete)
  #correct) on behavioral tasks which examine Negative Emotionality (Emotional go/nogo) and subscale and total scale scores on self-report measures of Negative Emotionality (Buss Perry Aggression)
Time Frame: 5 hours
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Self-report on Measure of Interoception Across Conditions
Description: Performance (time to complete)
Time Frame: 5 hours
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Self-report on Measure of Metacognition Across Conditions
Description: Performance (time to complete)
Time Frame: 5 hours
Reporting Status: Not Posted

9. Other Pre Specified Outcome: Self-report on Measure of Sleep Quality Across Conditions
Description: Performance (time to complete)
Time Frame: 5 hours
Reporting Status: Not Posted

10. Other Pre Specified Outcome: Between-group Differences in Brain Connectivity as Measured by Spectral Dynamic Causal Modeling (DCM) and Deterministic Dynamic Causal Modeling
Description: Between-group differences in brain connectivity as measured by Spectral dynamic causal modeling (DCM) and Deterministic dynamic causal modeling
Time Frame: 1 month
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: 1 month
Description: AE form/log
Arm/Group | Individuals With Cocaine Use Disorder | Individuals With Opioid Use Disorder | Individuals With Marijuana Use Disorder | Healthy Controls
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/97 | 0/51 | 0/108
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/97 | 0/51 | 0/108
Other Adverse Events (participants affected / at risk) | 0/50 | 0/97 | 0/51 | 0/108
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Individuals With Cocaine Use Disorder (N=50) | Individuals With Opioid Use Disorder (N=97) | Individuals With Marijuana Use Disorder (N=51) | Healthy Controls (N=108)
hospitalization (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0) — Participant was hospitalized to treat cellulitis of a vein that occurred as a result of plasma donation the day prior to study enrollment.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-06-12): https://cdn.clinicaltrials.gov/large-docs/69/NCT03495869/Prot_SAP_001.pdf
  • Informed Consent Form (2019-11-22): https://cdn.clinicaltrials.gov/large-docs/69/NCT03495869/ICF_000.pdf